CLINICAL TRIAL: NCT05605665
Title: Therapeutic Effect of Low Dose IL-2 Combined With Rapamycin in on sjögren's Syndrome
Brief Title: Low-dose Interleukin-2 and Rapamycin on sjögren's Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rapa-IL2-SS
Record Dates: First submitted 2022-10-29; First posted 2022-11-04 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Sjögren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Interleukin-2; aldesleukin; Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose interleukin-2 (Active Comparator): One million IU of IL-2 was injected subcutaneously once twice a week for 12 weeks.
  Interventions: Drug: low-dose interleukin-2
- Rapamycin (Active Comparator): Rapamycin 0.5ml once per day for 12 weeks.
  Interventions: Drug: rapamycin
- Low-dose interleukin-2 and rapamycin (Experimental): One million IU of IL-2 was injected subcutaneously twice a week and rapamycin 0.5ml once per day for 12 weeks.
  Interventions: Drug: low-dose interleukin-2; Drug: rapamycin

INTERVENTIONS:
Drug: low-dose interleukin-2 — low dose interleukin-2 injected subcutaneously, at a dose of 1 x 10~6 IU once twice a week, for 12 weeks.
  Other Names: Recombinant Human Interleukin-2
  Arms: Low-dose interleukin-2; Low-dose interleukin-2 and rapamycin
Drug: rapamycin — Rapamycin 0.5ml was taken orally once per day
  Other Names: sirolimus
  Arms: Low-dose interleukin-2 and rapamycin; Rapamycin

SUMMARY:
The purpose of this paper is to analysis of therapeutic effect and immunological mechanism of low-dose IL-2 combined with rapamycin in the treatment of Sjogren's syndrome

DETAILED DESCRIPTION:
A randomized, open clinical trial was designed. Patients will be randomly divided into three groups，including Ld-IL2 group, rapamycin group, Ld-IL2+rapamycin group. The improvement of clinical and laboratory indexes will be evaluated. Changes of immune cell subsets and cytokines will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, and aged 18-70 at the time of screening visit.
2. Patients with Sjogren's syndrome who meet the 2002 EULAR classification criteria.
3. If the standardized treatment is not effective or relapses, it is clinically necessary to give additional immunomodulatory treatment.
4. Disease activity: ESSDAI≥4 points.
5. The pregnancy test results of female subjects of childbearing age should be negative at screening and baseline.
6. The written informed consent form approved by the Ethics Committee of Peking University People's Hospital was signed and dated by the subject or legal representative.

Exclusion Criteria:

1. Severe chronic liver, kidney and heart dysfunction.
2. Severe drug-resistant bacterial infections, such as bacteremia and septicemia.
3. Patients with tumor and tumor history.
4. Chronic respiratory failure.
5. Patients who are ineffective in high-dose hormone pulse therapy.
6. Those who use rituximab or other biological agents within 3 months.
7. Patients with active tuberculosis infection or potential tuberculosis infection.
8. There are obstacles that can't cooperate or cause interference in completing this research: such as mental patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of Treg cells in peripheral blood | week 12
  Proportion of Treg cells in peripheral blood will be detected by flowcytometry

SECONDARY OUTCOMES:
ESSDAI [potential score 0 - 123] | week 12
  ESSDAI is [European League Against Rheumatism (EULAR) Sjögrens Syndrome Disease Activity Index]. Higher scores mean a worse outcome.
Physician's Global Disease Activity VAS, (potential score 0 - 10) | week 12
  Physician's Global Disease Activity (10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the myositis). Higher scores mean a worse outcome.
Patient's Global Disease Activity VAS, (potential score 0 - 80) | week 12
  Patient's Global Disease Activity (10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the myositis). Higher scores mean a worse outcome.
Rate of Participants with adverse effects associated with experimental drugs | week 12
  Adverse effects include fever, rash, abnormal liver function, rate of new-onset infection and any abnormal measures associated with low-dose IL-2 therapy, and oral ulcer, rash, hypertension, anemia, arthralgia, diarrhea and any abnormal measures associated with rapamycin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Study Director — Peking university peoples hospital
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China